CLINICAL TRIAL: NCT02057523
Title: Acthar as Rescue Therapy for Transplant Glomerulopathy in Kidney Transplant Recipients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to enroll patients, no longer at institution.
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Sanjeev Akkina, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0764
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Proteinuria; Transplant Glomerulopathy
MeSH Terms: conditions — Proteinuria | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acthar (Experimental): Acthar 80 units twice weekly for 6 months. If endpoint is not reached, duration may be increased to 12 months.
  Interventions: Drug: Acthar

INTERVENTIONS:
Drug: Acthar — Those interested will be started on Acthar 80 units twice weekly for 6 months. Those with minor adverse effects such as weight gain, worsening hypertension, or glucose intolerance will have their doses reduced to 40 unit twice weekly. Those with major adverse effects such as allergy or infection will discontinue the medication. If the primary endpoint of 50% reduction in proteinuria or total proteinuria less than 150mg/day is not reached, therapy may be continued for a total of 12 months.
  Other Names: Repository Corticotropin Hormone; Acthar Gel; Adrenocorticotropic Hormone

SUMMARY:
The goal of this study is to evaluate the benefit of ACTH (Acthar) in reducing proteinuria associated with transplant glomerulopathy in non-diabetic kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients with confirmed transplant glomerulopathy on kidney biopsy.
* Failed standard therapy (>25% reduction in proteinuria) including maximum use of an ACE inhibitor, ARB, or aldosterone blocker with a goal blood pressure less than 130/80 and optimization of their immunosuppression

Exclusion Criteria:

* Diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Akkina, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acthar
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Acthar
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: 50% Reduction in Proteinuria or Proteinuria < 150mg/Day
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: 25% Improvement in the MDRD eGFR
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Acthar
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No